CLINICAL TRIAL: NCT06342479
Title: The Effect of Discharge Training Given to Patients Having Intertrochanteric Fracture Surgery on Discharge Readiness and Surgical Recovery
Brief Title: Discharge Training for Patients With Intertrochanteric Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Yasemin Erden, Principal Investigator, Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NM: 04.20.ND:30.03.2023
Record Dates: First submitted 2024-03-20; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discharge training given (Experimental): In addition to the standard clinical monitoring applied in the clinic in a quiet and calm environment in the patient's room, outside of the doctor's visit, meal time, visiting and treatment hours and approximately two hours after the painkiller application, approximately 30 minutes (related to the subjects included in the developed booklet, nutrition, Discharge training (such as surgical recovery, movement, excretion, self-care skills, pain, exercise) will be given to patients. The patient will be asked to demonstrate the trainings (movements, exercises, etc.) that are explained to the patient by doing them at least three times. At the end of the training, a booklet prepared in accordance with the surgery the patient underwent will be given to the patient.
  Interventions: Behavioral: Discharge Education
- No discharge training provided (No Intervention): Patients included in the control group will receive routine discharge training and clinical follow-up at the Orthopedics Clinic. During standard clinical follow-up, service nurses provide verbal information to patients hospitalized in the Orthopedic Clinic about wound care, signs of infection at the wound site, medication use and post-discharge control times before discharge, but no written training materials are used.

INTERVENTIONS:
Behavioral: Discharge Education — Discharge education will be provided.
  Arms: Discharge training given

SUMMARY:
This study examines the effect of discharge training given to patients with intertrochanteric femur fractures on the wound healing process and readiness for discharge. In the study, patients were provided with certain educational content before and after discharge. The effect of training on wound healing, readiness for discharge and post-discharge recovery process will be evaluated statistically.

DETAILED DESCRIPTION:
Purpose of the study: This study will be conducted to determine whether the discharge training given to patients who underwent intertrochanteric femur fracture surgery has an effect on surgical recovery and readiness for discharge. The research is prospective and aimed to be a case-control group. The universe of the research; It will consist of patients hospitalized in the orthopedics service of Elazığ Fethi Sekin City Hospital and Fırat University Faculty of Medicine Research Hospital. The sample is; With the power analysis, 60 patients will constitute the population with a 0.05 error, 0.95 confidence interval, 0.6 effect size, and a representative power of 0.80. (n=60) Patients will be divided into 30 intervention groups and 30 control groups. Sociodemographic form, Toronto Wound Symptom Evaluation System Discharge readiness scale and patient evaluation form The data of the research will be collected using. Since the scales are publicly available, no permission will be sought from the authors. The research will be conducted with 60 patients who were hospitalized in the orthopedic clinic and underwent intertrochanteric femur fracture surgery. Groups will be divided into 30 intervention and 30 control groups. In order to prevent patients from interacting with each other during repeated measurements within the institution, 30 people were first admitted to the hospital. Control group; The next 30 people will constitute the intervention group patients.

* Type of research: The research is prospective and aimed to be a case-control group.
* Research questions/hypotheses:

  * What are the socio-demographic characteristics of the participants?
  * Does the discharge training given to participants have an effect on surgical recovery?
  * Is there any difference in surgical recovery according to the socio-demographic characteristics of the participants?
* Population-sample: The universe of the research; It will consist of patients hospitalized in the orthopedics service of Elazığ Fethi Sekin City Hospital and Fırat University Faculty of Medicine Research Hospital. The sample is; With the power analysis, 60 patients will constitute the population with a 0.05 error, 0.95 confidence interval, 0.6 effect size, and a representative power of 0.80. (n=60) Patients will be divided into 30 intervention groups and 30 control groups.

It is aimed to collect data face to face after obtaining ethics committee permission and institutional permission, and obtaining the necessary permissions from Elazığ Fethi Sekin City Hospital and Fırat University Faculty of Medicine Research Hospital. Before filling out the survey form, you will be informed about the research and a voluntary consent form will be read. All patients who agree will be included in the study. The research is aimed to be conducted between April 1 and December 1, 2023. All this operation will be carried out in accordance with the Declaration of Helsinki.

* Data collection tools: Sociodemographic form, Toronto Wound Symptom Evaluation System Discharge readiness scale and patient evaluation form The data of the research will be collected using. Since the scales are publicly available, no permission will be sought from the authors.
* How data will be collected: The research will be conducted with 60 patients who were hospitalized in the orthopedic clinic and underwent intertrochanteric femur fracture surgery. Groups will be divided into 30 intervention and 30 control groups. In order to prevent patients from interacting with each other during repeated measurements within the institution, 30 people were first admitted to the hospital. Control group; The next 30 people will constitute the intervention group patients.

After the patients included in the intervention group were evaluated in terms of the study participation criteria, they were informed by the researcher about the purpose, expected benefits and method of the study; Verbal and written informed consent forms will be obtained. The patient, for whom an informed consent form is obtained before discharge, will be evaluated for surgical recovery before discharge training is given. After the first evaluation, the standard clinical monitoring applied in the clinic in a quiet and calm environment in the patient's room, outside the doctor's visit, meal time, visiting and treatment hours, and approximately two hours after the painkiller application, in addition to the standard clinical monitoring, which takes approximately 30 minutes (with the topics in the developed booklet). Patients will be given discharge training (such as nutrition, surgical recovery, movement, excretion, self-care skills, pain, exercise). The patient will be asked to demonstrate the trainings (movements, exercises, etc.) that are explained to the patient by doing them at least three times. At the end of the training, a booklet prepared in accordance with the surgery the patient underwent will be given to the patient. Before the face-to-face interview with the patient is terminated, a telephone number will be obtained from the patient so that the evaluations can be made in the second, fourth and eighth weeks. In the second week after discharge, the researcher will call the patient from the phone number given by the patient and the questions in the section of the patient follow-up form created for the second week will be asked to the patient. The patient evaluation form will continue to be applied in the fourth and eighth weeks, as in the second week. When ending each phone call with the patient, information will be given about the time of the next phone call. Phone calls are planned to last approximately 10 minutes. In the second, fourth and eighth weeks after discharge, the application will continue as in the intervention group. After the study is completed, the developed discharge training booklets will be delivered to the control group patients.

* Evaluation of data: Data will be recorded and analyzed using the SPSS statistical package program.
* Difficulties and limitations of the research: The person may want to leave the study at a later time without stating any reason. Since the study is planned prospectively, the person may leave the study due to death or change of province.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish,
* At least primary school graduate,
* Patients who underwent intertrochanteric femur fracture surgery,
* Patients aged 18 and over will be included in the study.

Exclusion Criteria:

* Those who have a physical disability (such as vision, hearing, mobility) that prevents them from taking care of themselves,
* Those who have been diagnosed with a psychiatric disease (Dementia, Alzheimer, etc.)
* Those who have previously received discharge training
* Patients who are illiterate will be excluded from discharge training.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Toronto Wound Symptom Assessment System | 6months
  The Toronto Wound Symptom Assessment System-TYSDS was developed to evaluate the symptoms of patients with chronic wounds in 2009. Toronto Wound Symptom Assessment System - TYSDS is a tool consisting of 10 questions and each question gives a total of 11 points between 0-10. 0 in each question means that the symptom is not observed, and 10 means that the symptom is seen very intensely. A minimum score of 0 and a maximum of 100 points are obtained from the scale, and increasing scores indicate that the wound symptoms are more intense.

SECONDARY OUTCOMES:
Discharge readiness scale | 6months
  The scale is a 10-point Likert type scale, and if the average score from the scale is between 9-10, you are very ready to be discharged; if it is 8-8.9, you are very ready; if it is between 7-7.9, you are moderately ready; if it is below 7, you are very ready to be discharged. It is considered low readiness. Cronbach's alpha value of the discharge readiness scale was found to be .75.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Erden, Study Director — 54 / 5.000 Çeviri sonuçları Çeviri sonucu Erzurum Technical University Faculty of Health Sciences
Locations (1):
- Erzurum Technical University Faculty of Health Sciences, Erzurum, Turkey (Türkiye)